CLINICAL TRIAL: NCT06699810
Title: Modeling Ketosis-Prone Diabetes Remission Via Diverse Mechanisms of Glucotoxicity
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Priyathama Vellanki, Associate Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00008366
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Ketosis Prone Diabetes
Keywords: diabetic ketoacidosis; type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetic Ketoacidosis; Diabetes Mellitus, Type 2 | interventions — Continuous Glucose Monitoring; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Continuous Glucose Monitoring with Adjusted Insulin Doses (Experimental): Patients with ketosis-prone diabetes will wear a continuous glucose monitor (CGM) from the time of hospital discharge until insulin discontinuation. Insulin doses will be adjusted based on CGM glucose readings.
  Interventions: Device: Continuous Glucose Monitoring; Drug: Insulin

INTERVENTIONS:
Device: Continuous Glucose Monitoring — After insulin discontinuation participants continue wearing their CGMs, for a total of 3 months.
  Other Names: Freestyle Libre
Drug: Insulin — Participants will receive standard-of-care insulin treatment. Insulin dosing will be adjusted based on CGM glucose readings.

SUMMARY:
The goal of this study is to quantify day-to-day changes in blood glucose during treatment towards remission in ketosis-prone diabetes (KPDM) and describe them using a mathematical model of KPDM pathogenesis and remission.

DETAILED DESCRIPTION:
Approximately half of newly diagnosed obese African Americans presenting with diabetic ketoacidosis (DKA) have clinical, metabolic and immunologic features of type 2 diabetes (T2D), also known as ketosis-prone diabetes (KPDM). Unlike patients with type 1 diabetes, with intensive insulin treatment, approximately 70% of patients with KPDM exhibit improved pancreatic β-cell function and insulin sensitivity to allow discontinuation of insulin therapy (indicating near-normoglycemia remission based on fasting blood glucose (FBG) < 130 mg/dl and HbA1c < 7% off insulin therapy during follow-up]). The clinical course of KPDM is variable, with the duration of remission ranging from 6 to 120 months. The origins of this variation in the ability to achieve remission and its duration are poorly understood.

It has been observed that a 20-hour infusion of glucose reduces pancreatic beta (β)-cell function in a KPDM patient, and ketotic relapse is often preceded by hyperglycemia. The researchers thus hypothesized that the differences between conventional T2D and KPDM may be explained by the presence of a reversible glucotoxicity process, which operates on the timescale of days. The researchers developed a preliminary mathematical model describing the pathogenesis and remission of KPDM using such a process. The researchers showed that, by changing the rate of this hypothesized glucotoxicity process, this model can produce a variety of clinical courses, describing both conventional T2D and KPDM with varying rates and durations of remission.

This study is a pilot study that will refine and validate this model using prospective clinical data with continuous glucose monitor (CGM) data from patients with KPDM.

Patients will receive standard-of-care treatment for their diabetes as per their treating physician. Insulin therapy is the standard of care after an episode of DKA. Therefore, all participants will be discharged on insulin. A CGM will be placed on these participants at discharge from the hospital until insulin discontinuation. Since many of these patients insulin needs decrease after discharge from the hospital, the study team will utilize CGM glucose readings to adjust insulin doses.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent
* Have a BMI ≥ 28 kg/m2
* Be of African American ancestry
* Meet diagnostic criteria for DKA. Diagnostic criteria for DKA will include a plasma glucose > 250 mg/dl, a venous pH < 7.30, a serum bicarbonate < 18 mmol/l, and serum ketones (beta-hydroxy butyrate) > 1.5 mmol/L.

Exclusion Criteria:

* Significant medical or surgical illness including but not limited to myocardial ischemia, congestive heart failure, chronic peripheral venous insufficiency, chronic renal insufficiency, liver insufficiency (serum transaminases 3 times the upper limit of normal) and acute or chronic infectious processes
* Have recognized uncontrolled endocrine disorders such as hypercortisolism, acromegaly, or hyperthyroidism
* Anemia (hemoglobin < 12.5 g/dL for men, <11.5 gm/dL for women), bleeding disorders, or abnormalities in coagulation studies
* Pregnant
* Diagnosis of diabetes > 90 days before the presentation of DKA
* Unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-01-23 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Quantify Changes in Blood Glucose | Up to 3 months
  The day-to-day changes in blood glucose in KPDM will be quantified using CGMs.
Development of Mathematical Models | Up to 3 months
  The study team will adapt and develop mathematical models to describe the course of KPDM remission in each individual patient, i.e. the entire range of variation within the group of 12 participants.

SECONDARY OUTCOMES:
Correlation of Fit With Model Parameters and Duration of Remission | Up to 3 months
  The study team will validate mathematical models to predict duration of remission.

CONTACTS AND LOCATIONS:
Overall Officials: Priyathama Vellanki, MD, MS, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No